CLINICAL TRIAL: NCT00767455
Title: Evaluation of the Cumulative Irritation Potential of 828 Ointment in a Population of Normal Healthy Subjects
Brief Title: Cumulative Irritation Potential of 828 Ointment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Healthpoint (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 828-101-09-010
Record Dates: First submitted 2008-10-04; First posted 2008-10-07 (Estimated); Results first posted 2014-03-14 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-01

CONDITIONS: Healthy Volunteers
Keywords: cumulative irritation; healthy adult volunteers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Positive, Negative Controls (Sham Comparator)
  Interventions: Device: HP828-101

INTERVENTIONS:
Device: HP828-101 — 21 day patches

SUMMARY:
Cumulative Irritation Patch Test

DETAILED DESCRIPTION:
Single site study that will evaluate the relative cumulative irritation potential of HP828-101 ointment compared to a negative control, Johnson's baby oil, and a positive control, 0.2% SLS v/v, following 21 daily applications to the skin of normal, healthy volunteers.

ELIGIBILITY:
1. SUBJECTS 1.1 SUBJECT POPULATION

Subjects will be normal, healthy volunteers of either gender aged 18 to 65 years.

Inclusion Criteria:

Subjects must satisfy all of the following criteria:

1. Subjects must be ambulatory, 18 to 65 years of age and in reasonably good health.
2. Subjects may be of any ethnicity or skin type provided their skin pigmentation does not interfere with evaluations.
3. Female subjects must be surgically sterile, post-menopausal or using an acceptable method of birth control and all females of childbirth potential must be willing to take a urine pregnancy test at the beginning and at the end of the study.
4. Minor deviations in normal medical history not considered to be clinically significant by the investigator and the sponsor will be permitted.
5. Subjects must refrain from sunbathing, using tanning salons, swimming or using hot tubs during the course of the study.
6. Bathing is permitted, however, subjects must agree to attempt to keep the patches as dry as possible.
7. Subjects must read and sign an IRB approved informed consent form.

Exclusion Criteria:

Subjects with any of the following conditions are not eligible for participation:

1. Any systemic disease or disorder, complicating factors or structural abnormality that would negatively affect the conduct or outcome of the study (i.e., hepatitis, acute or chronic renal insufficiency).
2. Use of a prescribed pain medication, prescribed or over-the-counter anti-inflammatory drugs, immunosuppressive drugs or prescribed antihistamine medication (steroid nose drops and/or eye drops are permitted). Use of any over-the-counter pain medication that is ingested in quantities exceeding label instructions.
3. Subjects who have received an investigational drug or have participated in a patch test within the past 28 days or who are currently participating in or plan to enter a clinical trial.
4. A history of non-compliance or subjects who are considered potentially unreliable.
5. A history of skin allergies, including known sensitivity or strong reactions to any cosmetics and/or personal care products, topically prepared medical dressings, tapes or adhesives.
6. A history of clinically significant skin diseases which may contraindicate participation, including psoriasis, active eczema, atopic dermatitis and active cancer, even if currently controlled through medication.
7. Current use of topical or oral antibiotics.
8. Use of topical medications at the test area 2 weeks prior to enrollment or any body lotions/oils/creams at the test area for 48 hours prior to enrollment and throughout the trial.
9. Female subjects who are pregnant, stop contraceptive measures, expect to become pregnant or who are breast-feeding.
10. Subjects with any condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
11. Subjects with hematological disorders or immunologic disorders (HIV positive, AIDS and Systemic Lupus Erythematosus).
12. Subjects with any significant organ abnormality or disorders including gastric ulcer/insulin dependent diabetes.
13. Subjects with any clinically significant illness (sought medical attention, fever, took prescription medication) within the 4 weeks prior to study entry.
14. History of asthma, chronic bronchitis or any other bronchospastic condition that requires medication.
15. Known history of either real or suspected allergy or sensitization to any test article ingredient.
16. Anticipated change in the use of a systemic medication during the study that may affect the conduct or outcome of the study. Subjects must be stabilized on these medications for at least one month prior to receiving study drug and continue the same regimen throughout the study.
17. Bilateral mastectomy involving removal of lymph nodes.
18. Treatment of any type of cancer within the last six months.
19. The Principal Investigator may declare any subject ineligible for a sound medical reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2008-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Chair — Healthpoint; Innes Cargill, PhD, Study Director — Healthpoint
Locations (1):
- RCTS, Inc., Irving, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers >= 18 years of age
Groups:
- HP828-101 vs. Negative Control vs. Positive Control: Each subject was their own control and received patches containing approximately 200 mg of all three (test article, negative control, and positive control)
Period: Overall Study
Arm/Group | HP828-101 vs. Negative Control vs. Positive Control
Started | 59
Completed | 40
Not Completed | 19
Not completed — Investigator error | 19

BASELINE CHARACTERISTICS:
Groups:
- HP828-101 vs. Negative Control vs. Positive Control: each subject was their own control and received patches of all (test article, negative control, and positive control)
Arm/Group | HP828-101 vs. Negative Control vs. Positive Control
Number analyzed (Participants) | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 58
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 59

OUTCOME MEASURES:

1. Primary Outcome: Presence of Cumulative Irritation
Description: Irritancy of each test article was evaluated by assessment of the application sites using the Berger and Bowman Scale. Observed responses (e.g., erythema and edema) were graded according to the protocol-specified grading scale [0 (no visible reaction) to 4 (severe erythema)] for each subject. The relative cumulative irritation potentials of the test article (HP828-101 Ointment) and the negative and positive controls were determined by summing the daily scores of the 21 days of testing; with an overall scale of 0 (no visible reaction from any subjects over the 21 days) to 3360 (severe erythema experienced by every subject over the 21 days).
Time Frame: 22 days
Population: Per protocol
Measure: Number; unit: units on a scale
Groups:
- HP828-101: Intervention test article
- Negative Control: Johnson's Baby Oil
- Positive Control: Sodium Lauryl Sulfate
Arm/Group | HP828-101 | Negative Control | Positive Control
Number analyzed (Participants) | 40 | 40 | 40
units on a scale | 163.0 | 109.0 | 2073.0

ADVERSE EVENTS:
Time Frame: 22 days
Arm/Group | HP828-101 vs. Negative Control vs. Positive Control
Serious Adverse Events (participants affected / at risk) | 0/59
Other Adverse Events (participants affected / at risk) | 4/59
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HP828-101 vs. Negative Control vs. Positive Control (N=59)
Tape Reaction (Skin and subcutaneous tissue disorders) | 4 (4) — None of the adverse events were related to the test article. The four (4) subjects with a moderate adverse event due to tape irritation were discontinued from the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less